CLINICAL TRIAL: NCT07028892
Title: Gamified Learning for Pressure Injury Prevention: A Randomized Controlled Trial to Enhance Knowledge, Skills, and Attitudes Among Nurses
Brief Title: Gamified Learning for Pressure Injury Prevention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Collaborators: University of Massachusetts Chan Medical School, Worcester (Unknown); Massachusetts College of Pharmacy and Health Science (Other)
Responsible Party: Principal Investigator, Sinan Aydoğan, Assistant Professor, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MehmetAkifU-SBF-SA-2; 40099 (Other Grant/Funding Number: American Association of Critical-Care Nurses)
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pressure Injuries; Pressure Ulcer Prevention
Keywords: intensive care nurses; gamification; mobile learning; pressure injuries
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group will receive an education about pressure injury prevention via a gamified mobile application
  Interventions: Device: A gamified mobile learning
- Control Group (Active Comparator): The Control Group will receive the training via a booklet.
  Interventions: Other: Booklet training

INTERVENTIONS:
Device: A gamified mobile learning — There will be a gamified environment in a mobile application with case scenarios on pressure injury prevention designed by researchers.
  Arms: Experimental Group
Other: Booklet training — Nurses will receive training via a booklet about prevention of pressure injuries.
  Arms: Control Group

SUMMARY:
The goal of this Randomized Controlled Trial is to define the effect of gamified teaching methods for pressure injury prevention in intensive care nurses. The main questions it aims to answer are:

H1: The gamified learning experience will increase the nurses' knowledge of pressure injury prevention compared to the control group.

H2: The gamified learning experience will increase the nurses' skills in pressure injury prevention compared to the control group.

H3: The gamified learning experience will increase the nurses' attitude toward pressure injury prevention compared to the control group.

Researchers will compare two arm to see if there is a difference in knowledge, skills, and attitudes. Participants in the experimental group will be educated via a gamified mobile learning application.

DETAILED DESCRIPTION:
The inclusion criteria for the participants are: (a) being a registered nurse for more than one year, (b) being more than 18 years old, (c) having at least an associate degree in nursing, and (d) having a smartphone or tablet to be able to download the game application.

The Pressure Ulcer Knowledge Assessment Tool (PUKAT) will assess PI knowledge (Manderlier et al., 2017)

The Attitude Towards Pressure Ulcer Prevention instrument (APuP) will assess PI attitude (Beeckman et al., 2010) .

PI assessment skills will be performed in the skills laboratory at the Tan Chingfen Graduate School of Nursing with pressure injuries in various stages (stage one, stage two, stage three, stage four, unstageable stage, and deep tissue pressure injury) on the wound model. The researchers will create and validate a "Pressure Injury Evaluation Form."

ELIGIBILITY:
Inclusion Criteria:

* Being Registered Nurse for more than 1 year
* Having at least an associate degree of nursing
* Having a smart-phone or tablet
* Being more than 18 years old

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Pressure Ulcer Knowledge Level | 10 weeks
  The Outcome will be measured by "The Pressure Ulcer Knowledge Assessment Tool (PUKAT 2.0)". PUKAT 2.0 is a 26-item questionnaire that assesses nurses' knowledge of pressure injury in six areas: etiology and development (six items), classification and observation (five items), risk assessment (two items), and nutrition (one item).
Attitude Towards Pressure Ulcer Prevention | 10 weeks
  Attitude Towards Pressure Ulcer Prevention instrument (APuP) will be used for defining attitude level of ICU nurses. APuP is a reliable and valid instrument to assess attitudes towards pressure ulcer prevention. There are 13 items in this scale, each of them evaluated with a 5-point Likert.

SECONDARY OUTCOMES:
System Usability | 10 weeks
  System Usability Scale (SUS) will be used. In this study, a gamified mobile application for the prevention of pressure injuries will be developed. SUS will be used to evaluate the usability of the application.

CONTACTS AND LOCATIONS:
Overall Officials: Semiha Asli Bozkurt, Ph.D., Principal Investigator — Massachusetts College of Pharmacy and Health Science
Locations (1):
- UMass Chan Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aydogan S, Caliskan N. A Descriptive Study of Turkish Intensive Care Nurses' Pressure Ulcer Prevention Knowledge, Attitudes, and Perceived Barriers to Care. Wound Manag Prev. 2019 Feb;65(2):39-47. PMID 30730304
- [Background] Bozkurt, S. A., Samia, R., & Gazarian, P. K. (2023). Using standardized patient simulation in undergraduate nursing education: A scoping review. Clinical Simulation in Nursing, 74, 3-18. https://doi.org/10.1016/j.ecns.2022.10.003
- [Background] Beeckman D, Defloor T, Demarre L, Van Hecke A, Vanderwee K. Pressure ulcers: development and psychometric evaluation of the attitude towards pressure ulcer prevention instrument (APuP). Int J Nurs Stud. 2010 Nov;47(11):1432-41. doi: 10.1016/j.ijnurstu.2010.04.004. Epub 2010 May 14. PMID 20466370
- [Background] Manderlier B, Van Damme N, Vanderwee K, Verhaeghe S, Van Hecke A, Beeckman D. Development and psychometric validation of PUKAT 2.0, a knowledge assessment tool for pressure ulcer prevention. Int Wound J. 2017 Dec;14(6):1041-1051. doi: 10.1111/iwj.12758. Epub 2017 May 26. PMID 28547752